CLINICAL TRIAL: NCT06227650
Title: Closed-loop Insulin Delivery Systems ("Artificial Pancreas") in Patients With Pancreatitis or Pancreatectomy-induced Diabetes: an Observational Case Series
Brief Title: Closed-loop Insulin Delivery Systems in Pancreatic Diabetes
Acronym: IADIASP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0057
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Secondary Pancreatic Diabetes
Keywords: Closed-loop insulin delivery systems; artificial pancreas; pancreatitis; pancreatectomy; secondary diabetes; continuous glucose monitoring
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group1: Patients with secondary pancreatic diabetes equipped with a hybrid closed loop insulin delivery device
  Interventions: Device: hybrid closed loop insulin delivery system

INTERVENTIONS:
Device: hybrid closed loop insulin delivery system — Patients with secondary pancreatic diabetes equipped with a hybrid closed loop insulin delivery device

SUMMARY:
The purpose of this study is to evaluate the metabolic and the safety outcomes in people living with pancreatic diabetes (pancreatitis or pancreatectomy-induced diabetes) and using a closed-loop insulin delivery systems ("artificial pancreas").

DETAILED DESCRIPTION:
Secondary pancreatic diabetes is an unstable diabetes, due to deficiency in B cells which produce insulin, alpha cells which produce glucagon, and exorcrine insufficiency. Patients with secondary pancreatic diabetes are exposed to high glycemic variability and severe hypoglycemic episodes. Hybrid closed loop treatment has shown efficacy and safety for patients with type 1 diabetes and has the potential to improve the control of secondary pancreatic diabetes but has rarely been studied in this particular indication.

A retrospective observational cohort study in patients will be contucted suffering from secondary pancreatic diabetes in whom this device was implemented in order to observe metabolic and safety outcomes compared to the period before they were treated with hybrid closed-loop system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Presenting secondary pancreatic diabetes
* Treatment with insulin closed-loop delivery

Exclusion Criteria:

* Patient who objected to the use of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with secondary pancreatic diabetes and implementation of automated insulin therapy in BF
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the target | at day 0
  Percentage of time spent in the target, between 70 and 180 mg/dl: 14 to 90 days before starting hybrid closed loop
Percentage of time spent in the target | at day 90
  Percentage of time spent in the target, between 70 and 180 mg/dl the last 90 days available (T1) after starting hybrid closed loop

SECONDARY OUTCOMES:
Percentage of time spent | at day 0
  Percentage of time spent bellow 70 mg/dL (TBR for Time Bellow Range ) and Above 180 mg/dL (TAR for Time Above Range )
Percentage of time spent | at day 90
  Percentage of time spent bellow 70 mg/dL (TBR for Time Bellow Range ) and Above 180 mg/dL (TAR for Time Above Range )
Pourcentage of closed-loop mode use | at day 90
  Pourcentage of closed-loop mode use
Hypoglycemia events (serveral hypoglycemia ) | at day 0
  Number of serveral hypoglycemia events requiring hospitilisation and/or emergency
Hypoglycemia events (serveral hypoglycemia ) | at day 90
  Number of serveral hypoglycemia events requiring hospitilisation and/or emergency
Hyperglycemia events | at day 0
  Number of hyperglycemia events requiring hospitalisation and /or emergency
Hyperglycemia events | at day 90
  Number of hyperglycemia events requiring hospitalisation and /or emergency
Glucose Management Indicator (GMI) | at day 0
  Glucose Management Indicator (GMI)
Glucose Management Indicator (GMI) | at day 90
  Glucose Management Indicator (GMI)
Coeffecient of variabilty of Glucose Management Indicator | at day 0
  Coeffecient of variabilty
Coeffecient of variabilty of Glucose Management Indicator | at day 90
  Coeffecient of variabilty
Microangiopathic events | at day 0
  Number of microangiopathic events (diabetic retinopathy ,diabetic nephropathy, diabetic neuropathy )
Microangiopathic events | at day 90
  Number of microangiopathic events (diabetic retinopathy ,diabetic nephropathy, diabetic neuropathy )

CONTACTS AND LOCATIONS:
Overall Officials: Alfred PENFORNIS, PHD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, Fra, France

IPD SHARING:
Plan to Share IPD: No